CLINICAL TRIAL: NCT07104682
Title: An Open Label Individual Patient Study Investigating the Safety and Efficacy of GCAR1 in a Patient With Metastatic Relapsed Alveolar Soft Part Sarcoma
Brief Title: A Study to Determine the Safety and Effectiveness of the Investigational Cellular Therapy GCAR1 in a Patient With Alveolar Soft Part Sarcoma
Acronym: CLIC-YYC-GPNMB
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HREBA.CC-25-0218
Record Dates: First submitted 2025-07-29; First posted 2025-08-05 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Alveolar Soft Part Sarcoma (ASPS); Sarcoma
MeSH Terms: conditions — Sarcoma, Alveolar Soft Part; Sarcoma

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GCAR1 (Experimental): The patient may receive two separate intravenous infusions of cryopreserved, autologous GCAR1, each containing a total of 5.0E6 CAR+ T cells/kg patient body weight. Both infusions will be preceded by standard lymphodepleting chemotherapy (Fludarabine 40 mg/m2 x 3 days, cyclophosphamide 600 mg/m2 x 2 days). The patient will only be eligible to receive a second dose if they had a partial response (PR), stable, or progressive disease (SD/PD) by RECIST 1.1 criteria after receiving Dose 1. A second infusion should not be administered if the patient achieves and sustains a complete response on disease assessment. Dose 2 will be administered at physician discretion and must be given at minimum 60 days and a maximum of 730 days post administration of Dose 1. For the patient to proceed with a second infusion, any toxicity that does not meet the criteria of a Dose Limiting Toxicity must be assessed for clinical significance, and taken into consideration by the PI before proceeding.
  Interventions: Biological: GCAR1

INTERVENTIONS:
Biological: GCAR1 — GCAR1 is a patient-specific cell therapy product containing a mixture of autologous lymphocytes transduced with a lentiviral vector encoding a chimeric antigen receptor (CAR) targeting GPNMB. The CAR comprises a single-chain variable fragment (scFv) binding domain derived from a fully human GPNMB-specific monoclonal antibody (CDX-011), a CD8 hinge and transmembrane domain, a myc sequence for product identification, and the CD137 (4-1BB) and CD3 zeta chain intracellular signaling domains. After infusion, the autologous GPNMB CAR T-cells expressing the genetically engineered anti-GPNMB CAR enable the specific targeting of GPNMB-expressing cells. Upon binding to GPNMB-expressing cells, the CAR transmits T cell activation signals that promote the elimination of target cells through CAR T cell degranulation and the release of cytotoxic molecules. The cellular signal also facilitates CAR T cell proliferation and persistence that may enable prolonged disease control through immunosurveillance

SUMMARY:
A single patient study to determine whether GCAR1 is safe and effective for refractory, progressive metastatic alveolar soft part sarcoma (ASPS).

DETAILED DESCRIPTION:
CLIC-YYC-GPNMB-05 is an Open Label Individual Patient (OLIP)/Single Patient Study (SPS) developed according to the Health Canada template and guidelines released in 2019 for studies to access therapies not otherwise available to patients, in the situation where there are no options of treatment or cure remaining. The patient under consideration for CLIC-YYC-GPNMB-05 has refractory, progressive metastatic alveolar soft part sarcoma (ASPS). There are no standard therapies for metastatic ASPS known to provide potential for cure, and there are no clinical trials available in Canada for consideration. We propose to treat the patient with GCAR1, a patient-specific cell therapy product containing a mixture of autologous lymphocytes transduced with a lentiviral vector containing a chimeric antigen receptor (CAR) that enables the specific targeting towards tumor cells expressing the cell surface protein glycoprotein non-metastatic B (GPNMB).

ELIGIBILITY:
Inclusion Criteria:

* The patient must have relapsed ASPS that is in the opinion of the treating physician not resectable, or that resection would be associated with significant morbidity.
* The patient must provide informed consent.
* The only other eligibility criteria is adequate organ function, defined as creatinine clearance >30 ml/min and LVEF >45%.

Exclusion Criteria:

* Any active uncontrolled infection
* Any anti-cancer therapy within 21 calendar days prior to the first dose of lymphodepleting chemotherapy

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Estimated)
Dates: Start 2025-08-08 (Estimated); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Treatment response | Diagnostic imaging (CT and/or MRI) will be performed at baseline (pre-treatment) and then subsequently at day 46 and day 91 after GCAR1 infusion, and at 6 months, 9 months and 12 months after last infusion to evaluate response to therapy.
  The overall response assessment considers the response of the target and non-target lesions and development of new lesions.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Calgary, Calgary, Canada